CLINICAL TRIAL: NCT05725070
Title: Phase 0/1 Theragnostic Study in Patients With Metastatic Castration Resistant Prostate Cancer in Need of Salvage Therapy, Selected by 18F-PSMA-PET Imaging and Treated by Alpha-therapeutic Radioligand 212Pb-NG001
Brief Title: Phase 0/1 Study of 212Pb-NG001 in mCRPC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ARTBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG001-01
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug (Experimental): 212Pb-NG001
  Interventions: Drug: 212Pb-NG001

INTERVENTIONS:
Drug: 212Pb-NG001 — 212Pb-NG001 is a targeted alpha-emitting radiopharmaceutical conjugated to a PSMA targeting peptide.
  Patients will receive an initial single 10 MBq dose IV to explore the imaging potential of 212Pb-NG001.

SUMMARY:
The purpose of this study is to evaluate the imaging feasibility and safety of 212Pb-NG001.

DETAILED DESCRIPTION:
This is a single site, open label, non-randomized, non-controlled intervention study with an initial microdosing run-in part (phase 0), followed by a conventional dose-escalation phase 1 part.

ELIGIBILITY:
Key Inclusion Criteria:

* ECOG performance status of 0 to 2
* Life expectancy >6 months
* Histological, pathological, and/or cytological confirmation of prostate cancer
* Metastatic castration resistant prostate cancer
* Failure of conventional treatment or such treatment not available/accepted by patient
* PSMA avid mCRPC lesions confirmed by PSMA PET/CT
* Adequate hematopoietic, kidney and liver function

Key Exclusion Criteria:

* Concurrent or other cancer diagnosis last two years, except for carcinoma in situ
* Concomitant diseases not compatible for radioactive therapy
* Previous PSMA-targeted radioligand therapy
* Concurrent serious (as determined by the Principal Investigator) medical conditions

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of SPECT/CT gamma camera imaging for uptake of 212Pb-NG001 | Up to 28 days
  To qualitatively determine whether 212Pb-NG001 can be used to produce images of sufficient clarity and sensitivity by SPECT/CT to confirm 212Pb-NG001 uptake and biodistribution.

SECONDARY OUTCOMES:
Safety and tolerability | Up to 28 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Body clearance | Up to 2 days
  To study body clearance of 212Pb-NG001 by gamma camera imaging and by sample and probe measurements.
Therapeutic effect on prostate cancer as indicated by decreasing serum PSA and/or ALP | Up to 28 days
  To explore any signals of therapeutic effects on the laboratory parameters: prostate specific antigen (PSA) and alkaline phosphatase (ALP)

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Berner, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway